CLINICAL TRIAL: NCT01198496
Title: Phase IV Study for Effect of Intensive Blood-Pressure Control Using Anti-hypertensive Agents in Essential Hypertension With History of Stroke
Brief Title: Recurrent Stroke Prevention Clinical Outcome Study
Acronym: RESPECTS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Biomedis International Ltd. (Other)
Responsible Party: Kazuyuki Shimada/Board chairperson, RESPECT Study Group
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RESPECT 1; UMIN000002851 (Registry Identifier: UMIN Clinical Trial Registry)
Record Dates: First submitted 2010-08-28; First posted 2010-09-10 (Estimated); Last update posted 2012-07-31 (Estimated); Status verified 2010-09

CONDITIONS: Hypertension; Stroke; Blood Pressure
Keywords: hypertension; stroke; blood pressure
MeSH Terms: conditions — Hypertension; Stroke | interventions — Losartan; Hydrochlorothiazide; Amlodipine; Spironolactone; candesartan cilexetil; Valsartan; Telmisartan; Olmesartan Medoxomil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Blood pressure (Experimental): The incidence of recurrent stroke will be lower in a strict BP control group having lower BP target: less than 120/80 mmHg* than in a standard BP control group having BP target less than 140/90 mmHg or less than 130/80 mmHg for current DM/CKD/old MI in patients with hypertension.
  * This study uses BP target: less than 120/80 mmHg that is sat up for this study rather than the BP target recommended in the Guidelines for the management of hypertension, Japanese Society of Hypertension 2009.
  * BP management is strongly recommended in patients with hypertension, DM, and/or CKD for prevention of recurrent stroke in the Japanese guidelines for the management of stroke 2009.
  Interventions: Drug: Losartan, Losartan and HCTZ, Amlodipine , Spironolactone

INTERVENTIONS:
Drug: Losartan, Losartan and HCTZ, Amlodipine , Spironolactone — <Study drugs and treatment steps> Step 1: Losartan 50 mg in principle (other ARB is usable) Step 2: Combination drug containing losartan 50 mg and hydrochlorothiazide 12.5 mg Step 3: Combination drug containing losartan 50mg and HCTZ 12.5mg + amlodipine 5 mg Step 4: Losartan 50 mg + combination drug containing losartan 50 mg and HCTZ 12.5 mg + amlodipine 5 mg Step 5: Losartan 50 mg + combination drug containing losartan 50 mg and HCTZ 12.5 mg + amlodipine 10 mg Step 6: Losartan 50 mg + combination drug containing losartan 50 mg and HCTZ 12.5 mg + amlodipine 10 mg + spironolactone 25 mg
  Other Names: candesartan cilexetil; valsartan; telmisartan; olmesartan medoxomil

SUMMARY:
1. Objectives and Hypothesis

   1. Objectives:

      This study evaluates whether strict BP management is useful for the prevention of recurrent stroke.

      Hypertensive patients with history of stroke are treated with stepwise multi-drug therapy to achieve stricter BP target <120/80 mmHg in the strict BP control group and less stricter BP target <140/90 mmHg or <130/80 mmHg for patients with current DM/CKD/MI in the standard BP control group. The participants under the BP treatment achieving their respective BP target will be followed for recurrence of stroke. The study continues until the number of patients with the first recurrent stroke reaches a total of 330 between the two groups. The occurrence rates of recurrent stroke will be compared between the two groups.
   2. Hypotheses The incidence of recurrent stroke will be lower in a strict BP control group having lower BP target: <120/80 mmHg* than in a standard BP control group having BP target <140/90 mmHg or <130/80 mmHg for current DM/CKD/MI in patients with hypertension.
2. Study design This will be a multicenter, randomized, open-label study. The study consists of a screening period, a titration period and a follow-up period. The screening period is a period between the date of consent and the enrollment date. Hypertensive patients with history of stroke are randomly assigned to either the strict BP control group having the target of <120/80 mmHg or the standard BP control group having the target of <140/90 mmHg without current DM, CKD or MI and <130/80 mmHg with current DM, CKD or MI. The titration period is the period finding a treatment which achieves target BP, and 24 weeks at maximum. Patients will be treated with stepwise multi-drug therapy using an angiotensin-receptor antagonist, diuretic, calcium channel blocker and aldosterone antagonist. The participants will be observed under the BP management for their respective BP target. The study will be continued until the number of patients with the first recurrent stroke reaches a total of 330 between two groups. The follow-up period will be 3 years.

The recurrent rates of stroke in both groups will be compared from various aspects, and strict BP management will be investigated on the usefulness in prevention of recurrent stroke.

DETAILED DESCRIPTION:
Rationale for Study Duration Predicting that strict BP control reduces the relative risk of recurrent stroke by 30% during the planned observation period of 3 years, the number of participants necessary to detect the recurrent stroke with rate of 2.5%/year and 7.5%/3 years is 2482 patients per group with a detection power of 90% and α-error of 0.05. A drop-out rate is estimated as 20%.

Therefore, the study will be continued for 3 years until a total of 330 patients with recurrent stroke in both groups are identified.

Rationale for Dosing Regimen One of ARB, losartan, is chosen for Step 1 therapy, because angiotensin II receptor blocker (ARB) is preferred as the first line of anti-hypertensives. Furthermore, a stepwise combination therapy of BP lowering drugs diuretic, hydrochlorothiazide, and calcium channel blocker, amlodipine, will be used, because the Japanese guidelines recommend the combination for BP control in prevention of recurrent stroke. (Step 2 to Step 5). Finally (as Step 6), a selective aldosterone antagonist, spironolactone, will be added for the treatment of with refractory hypertensive patients whose BP does not reach to the target.

Treatment Plan The dosages of study drugs will be determined according to the package insert for the drug.

Patients who are not treated with antihypertensive agent or treated with one antihypertensive agent at enrollment will start from Step 1. Patients who are treated with two antihypertensive agents at enrollment will start from Step 2.

In principle, treatment duration will be for 4 weeks at each step.

ELIGIBILITY:
Inclusion Criteria:

Participants include those with essential hypertension and history of stroke who satisfy the following criteria:

* Outpatient
* Onset of stroke(cerebral infarction/cerebral hemorrhage) occurred between 30 days and 3 years prior to the date of consent.
* Drug adherence is ≧80% during the screening period.
* Mean of 2 baseline BP measurements(measured at outpatient clinic) within 30 days prior to the date of consent is either 180 >SBP ≧130 mmHg or 110 >DBP ≧80 mmHg (untreated -3 anti hypertensive agents patients).
* Cerebral infarction with severity 3 or less in the modified Rankin scale.

Exclusion Criteria:

Patient who meets any one of the following criteria is excluded from the study.

* Women who are pregnant, are possible pregnant, or are breastfeeding
* Possible secondary hypertension
* Severe hypertension (grade III or greater) with baseline SBP ≧180 mmHg or DBP ≧110 mmHg)
* Myocardial infarction or undergoing angioplasty occurred within 3 months prior to the screening.
* Current or previous heart failure with NYHA classification class III or more, or EF less than 35%
* Severe bilateral carotid stenosis or major cerebral artery occlusion
* Severe paralysis due to stroke (modified Rankin scale ≧ 4 )
* Current renal dysfunction (serum Cr ≧ 2.0 mg/dL right before the date of consent)
* Current hepatic dysfunction with AST or ALT value ≧ 100 IU/mL right before the date of consent
* Refractory hypertension treated with four or more antihypertensive drugs
* Hypersensitivity or allergy to losartan and other angiotensin II receptor blockers, hydrochlorothiazide, amlodipine or sulfonamide derivative
* Major surgery planned during the study period
* Participants of other clinical studies within the last 30 days
* Current malignancy (previous malignancy within 5 years after the end of treatment) excluding squamous-cell skin cancer
* Previous and current subarachnoid hemorrhage
* Definitive dementia 12) (based on a clinical diagnosis)
* Patients who have difficulty in signing consent or who do not agree to the provided consent
* Patients who are judged to be unsuitable for participating the study by the primary investigator or sub-investigator.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5000 (Estimated)
Dates: Start 2010-10; Primary Completion 2017-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
the prevention of recurrent stroke. | Until the first recurrent stroke reaches a total of 339 between the two groups
  Hypertensive patients with history of stroke are treated with stepwise multi-drug therapy to achieve BP target less than 120/80 mmHg in the strict BP group and BP target less than 140/90 mmHg or less than 130/80 mmHg for patients with DM/CKD/old MI in the standard BP group. The participants under the BP treatment achieving their respective BP target will be followed for recurrence of stroke. The study continues until the number of patients with the first recurrent stroke reaches a total of 339 between the two groups.

SECONDARY OUTCOMES:
The incidence of events other than stroke | Until the first recurrent stroke reaches a total of 339 between the two groups
  Under the strict BP control, not only the recurrence of stroke but also occurrence of cardiovascular events (such as myocardial infarction and heart failure), angioplasty, and death will be reduced.
  Separate hypothesis: Additionally, occurrence and exacerbation of dementia is also decreased under the strict BP control in comparison with the standard control.

CONTACTS AND LOCATIONS:
Overall Officials: Kazuyuki Shimada, MD, Study Chair — RESPECT Study Group
Locations (1):
- Jichi Medical Univercity, Shimotsuke, Tochigi, Japan

REFERENCES:
- [Derived] Saiz LC, Gorricho J, Garjon J, Celaya MC, Erviti J, Leache L. Blood pressure targets for the treatment of people with hypertension and cardiovascular disease. Cochrane Database Syst Rev. 2022 Nov 18;11(11):CD010315. doi: 10.1002/14651858.CD010315.pub5. PMID 36398903
- [Derived] Saiz LC, Gorricho J, Garjon J, Celaya MC, Erviti J, Leache L. Blood pressure targets for the treatment of people with hypertension and cardiovascular disease. Cochrane Database Syst Rev. 2020 Sep 9;9(9):CD010315. doi: 10.1002/14651858.CD010315.pub4. PMID 32905623
- [Derived] Kitagawa K, Yamamoto Y, Arima H, Maeda T, Sunami N, Kanzawa T, Eguchi K, Kamiyama K, Minematsu K, Ueda S, Rakugi H, Ohya Y, Kohro T, Yonemoto K, Okada Y, Higaki J, Tanahashi N, Kimura G, Umemura S, Matsumoto M, Shimamoto K, Ito S, Saruta T, Shimada K; Recurrent Stroke Prevention Clinical Outcome (RESPECT) Study Group. Effect of Standard vs Intensive Blood Pressure Control on the Risk of Recurrent Stroke: A Randomized Clinical Trial and Meta-analysis. JAMA Neurol. 2019 Nov 1;76(11):1309-1318. doi: 10.1001/jamaneurol.2019.2167. PMID 31355878
- See also: RESPECT Study — http://www.respect-study.com